CLINICAL TRIAL: NCT05168904
Title: A Phase 1/2, Open Label, Multicenter Study to Investigate the Safety and Efficacy of Fadraciclib (CYC065), an Oral CDK 2/9 Inhibitor, in Subjects With Leukemias or Myelodysplastic Syndrome (MDS)
Brief Title: A Study to Investigate Fadraciclib (CYC065), in Subjects With Leukemia or Myelodysplastic Syndrome (MDS)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow enrollment and financial limitations
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYC065-102
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Leukemia; Myelodysplastic Syndrome(MDS)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — CYC065

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I Dose escalation (Experimental): Phase 1 = fadraciclib administered orally in escalating doses starting at 50mg bid MWF for 3 weeks of a 4-week cycle. Subsequent cohorts will escalate in dose and schedule until optimized phase 2 dose and schedule is achieved.
  Interventions: Drug: fadraciclib
- Phase 2 (Experimental): Recommended fadraciclib phase 2 dose and schedule administered orally in 28-day cycles.
  Interventions: Drug: fadraciclib

INTERVENTIONS:
Drug: fadraciclib — Fadraciclib is a highly selective, orally- and intravenously- available, 2nd generation amino-purine inhibitor of CDK2 and CDK9.
  Other Names: CYC065

SUMMARY:
This is a 2-part, phase 1/2, open-label, multicenter study designed to evaluate the safety and efficacy of fadraciclib (formerly CYC065) administered orally BID. This study consists of Phase 1 and Phase 2 components in subjects with Leukemia or Myelodysplastic syndrome (MDS) who have progressed despite having standard therapy or for which no standard therapy exists.

DETAILED DESCRIPTION:
Phase 1 part of the study will consist of a dose-escalation and a dose-finding component.

Phase 2 will enroll subjects AML, CLL, or MDS, into 7 groups:

Group 1: Subjects with AML or MDS having marrow blasts over > 10%, who have experienced an inadequate response or progression on venetoclax combinations with either HMAs or low dose Ara-C or similar venetoclax combinations

Group 2: Fadraciclib: Subjects with AML or MDS relapsed/refractory having marrow blasts over > 10% with FLT3, KIT, MAPK pathway (N and K RAS, BRAF, PTPN11, NF1) mutations after at least 1 line of prior therapy.

Group 3: Fadraciclib: Subjects with CLL who have progressed on 2 or more lines of therapy, including a Bruton's tyrosine kinase (BTK) inhibitor and venetoclax.

Group 4: Fadraciclib plus azacitidine: Subjects with AML or MDS who have progressed after therapy with an HMA.

Group 5: Fadraciclib plus venetoclax: Subjects with AML or MDS who have progressed after therapy with venetoclax.

Group 6: Fadraciclib plus venetoclax: Subjects with CLL or small lymphocytic lymphoma (SLL) who have progressed after therapy with venetoclax.

Group 7: Basket cohort: Leukemia types suspected to have a related mechanism of action such as MCL1, or MYC amplification/over-expression not included in previous groups

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years.
2. a) AML/MDS with blasts > 10% in subjects who have had an inadequate response or progression to venetoclax combinations with either HMA or low dose Ara-C or similar venetoclax combinations. or b. CLL in subjects who have received at least 2 lines of therapy, including venetoclax and a BTK inhibitor, who require therapy as per iwCLL criteria.
3. Any prior therapy must have been completed at least 2 weeks prior to enrollment on this protocol, and the participant must have recovered to eligibility levels from prior toxicity
4. Hydroxyurea may be used for the first 14 days of Cycle 1 for peripheral blast control. Valproic acid not being used for seizure control should be stopped 72 hours before starting treatment with fadraciclib.
5. Any prior therapy with decitabine or azacitidine must have been completed at least 3 weeks prior to enrollment on this protocol.
6. Subjects who relapsed post-autologous or post-allogeneic transplant are eligible. Post-transplant subjects must be without active fungal disease or significant acute graft-versus-host disease.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Women of childbearing potential (WOCBP) must have a negative pregnancy test (urine or serum) within 7 days prior to starting the study drug. Both males and females must agree to use effective birth control during the study (prior to receiving the first dose and for 6 months after the last dose) if conception is possible during this interval.
9. Subjects must be able to swallow and retain orally administered medication and not have any clinically significant GI abnormalities that may alter the absorption, such as malabsorption syndrome or major resection of the stomach or bowels.
10. Subjects must be able to agree to and sign the informed consent and to comply with the protocol.

Exclusion Criteria:

1. Subjects with known active leptomeningeal involvement by AML.
2. Subjects who have not received vaccines for SARS-COV-2 within the last 3 months and have suspected signs and symptoms of COVID-19 or a recent history (within 14 days) of contact with any COVID-19 positive subject/isolation/quarantine or subjects with confirmed COVID-19.
3. Subjects with a history of another primary malignancy, other than:

   1. Carcinomas in situ, e.g., breast, cervix, and prostate
   2. Locally excised non-melanoma skin cancer
   3. No evidence of disease from another primary cancer for 2 or more years and has not taken any anticancer treatment in 2 years.
4. Any other clinically significant acute or chronic medical or psychiatric condition or any laboratory abnormality that may increase the risk associated with study drug administration or may interfere with the interpretation of study results.
5. Diseases that significantly affect GI absorption of fadraciclib.
6. Subjects who have impaired cardiac function or clinically significant cardiac disease.
7. Presence of active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment.
8. Presence of an active infection requiring IV antibiotics.
9. Presence of known history of human immunodeficiency virus-1/2 with uncontrolled viral load and on medications that may interfere with metabolism.
10. Presence of active hepatitis B virus (HBV) or hepatitis C virus (HCV).
11. Subject has received systemic anticancer therapy (including investigational therapy), radiotherapy, or immunotherapy < 14 days or 5 half-lives (whichever is shorter) prior to administration of Dose 1 of study drug on Day 1 or have not recovered from the side effects of such therapy.
12. Major surgery/surgical therapy for any cause within 4 weeks of the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 months
  The incidence rate of dose-limiting toxicities (first cycle only) at each dose level
Overall Response Rate (ORR) | 18 months
  Assessment of response criteria according to iwCLL criteria for CLL/SLL and IWG criteria for AML and MDS.

SECONDARY OUTCOMES:
Adverse events | 24 months
  Type, frequency, and severity of adverse drug reactions

OTHER OUTCOMES:
Pharmacodynamics | 6 months
  To investigate CDK9-dependent transcription inhibition as assessed by differential target gene expression relative to baseline.
Pharmacogenomics | 24 months
  To investigate plasma cell-free DNA mutation and copy number variation profile of fadraciclib as determined by NGS.
Correlative studies | 24 months
  To investigate effect on epigenetics, immunomodulation and apoptotic pathway

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No